CLINICAL TRIAL: NCT00905463
Title: Analysis of Prognosis and Patient Reported Outcomes in Lung Transplant Candidates
Brief Title: Prognosis of Lung Transplant Candidates
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kyoto University, Graduate School of Medicine (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Responsible Party: Principal Investigator, Toru Oga, Respiratory Care and Sleep Control Medicine, Kyoto University, Graduate School of Medicine, Kyoto University, Graduate School of Medicine
Other Study IDs: E554kyoto
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Lung Transplantation; Respiratory Failure
Keywords: Lung transplant candidates; Health-related quality of life; patient reported outcome; Prognosis
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Lung Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Transplantation: Lung transplantation candidates
  Interventions: Procedure: Lung transplantation

INTERVENTIONS:
Procedure: Lung transplantation — Lung transplantation

SUMMARY:
The purposes of the study are (1) to analyze the baseline patient characteristics cross-sectionally, (2) to analyze the prognosis and its predictive factors and (3) to examine the longitudinal clinical course in the lung transplant candidates in Japan.

DETAILED DESCRIPTION:
The significance of assessing patient reported measurements including health status, dyspnea and psychological status has not been well investigated in the lung transplant candidates. Therefore, in the present study, we aim to examine (1) contributive factors to their health status based on baseline data, (2) whether patient reported measurements would predict patients' prognosis and (3) how they would change for 5 years as compared to physiological measurements.

ELIGIBILITY:
Inclusion Criteria:

* New lung transplant candidates

Exclusion Criteria:

* Heart and lung transplant candidates
* Uncontrolled severe comorbidities

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: University hospital clinic for lung transplantation
Sampling Method: Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2009-04; Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Prognosis/Mortality | 5 years

SECONDARY OUTCOMES:
Health status | At entry and every year for 5 years
Dyspnea | At entry and every year for 5 years
Psychological status | At entry and every year for 5 years
Sleep quality | At entry and every year for 5 years
Pulmonary function | At entry and every year for 5 years
Arterial blood gas | At entry and every year for 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Date, MD, PhD, Study Chair — Graduate School of Medicine, Kyoto University
Locations (4):
- Japan (4):
  - Graduate School of Medicine, Kyoto University, Kyoto
  - Okayama University, Okayama
  - Tohoku University, Sendai
  - Osaka University, Suita